CLINICAL TRIAL: NCT01832415
Title: Non Interventional Study Dealing With the Use of Bevacizumab (Avastin®) in Patients With Epithelial Ovarian Cancer, Fallopian Tube or Primary Peritoneal and Treated in First-line Therapy
Brief Title: First Line Ovarian Cancer Treatment - Cohort Study
Acronym: ENCOURAGE
Status: Completed | Type: Observational
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ENCOURAGE (GINECO-OV123)
Record Dates: First submitted 2013-03-28; First posted 2013-04-16 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Epithelial Ovarian Cancer
Keywords: First line treatment; Ovarian cancer; Avastin; fallopian tube or primary peritoneal
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Use of bevacizumab (Avastin ®) - First-line ovarian cancer: Patient receiving bevacizumab in ovarian cancer first line treatment
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Observation of bevacizumab administration in first line ovarian cancer treatment

SUMMARY:
The French cooperative group GINECO proposes to implement an observational study to describe a real situation, in daily practice tolerance and methods of administration of bevacizumab (Avastin ®)

DETAILED DESCRIPTION:
Population: Patients aged 18 years and older with an epithelial ovarian cancer, fallopian tube or primary peritoneal or witch it was decided to initiate a process comprising of Bevacizumab (Avastin ®) in first-line therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over,
* Patients with an epithelial ovarian cancer, fallopian tube or peritoneal who will receive bevacizumab (Avastin ®) in first-line therapy
* Patients should be informed of the study orally and should not have any objection their data to be processed.

Exclusion Criteria:

* Patient participation in a clinical trial
* Patient non-affiliated to a social security scheme.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Patients with epithelial ovarian cancer, fallopian tube or peritoneal with treatment receiving Bevacizumab (Avastin ®) in first-line therapy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety according to CTCAE v4.0 criteria | Patient will be followed dureing 36 months
  To assess patient safety and the tolerance of bevacizumab andministered regarding the daily practice of the oncologist.

SECONDARY OUTCOMES:
Efficacy | Patient will be followed during 36 months
  • Evaluate the efficacy of bevacizumab (Avastin ®) in terms of progression-free survival (PFS) .
Efficacy of treatment at relapse | Patient will be followed during 36 months
  Evaluate the efficacy of the treatment that will be administered at the disease relapse.
Characteristics of the population registered | At registration
  Discribe the population that will be registered to make correlation with the safety and efficacy measure
Indication and cons indication of bevacizumab in clinical practice | At registration
  Discribe the reason why patient receive or not bevacizumab in first line of ovarian cancer treatment
Evaluation of monitoring practices of bevacizumab | The patients will be followed during 36 months
  Discribe the method that are used during a treatment by bevacizumab in the daily practice
Evaluation of the modality of use of bevacizumab | The patients will be followed during 36 months
  Discribe how bevacizumab is administered in the daily practice

CONTACTS AND LOCATIONS:
Overall Officials: Dominique BERTON-RIGAUD, MD, Principal Investigator — ICO de l'Ouest, Site René Gauducheau - Saint-Herblain
Locations (14):
- France (14):
  - Centre Paul Papin, Angers
  - Clinique Tivoli, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Intercommunal, Fréjus
  - institut Paoli Calmette, Marseille
  - Clinique Valdegour, Nîmes
  - Centre Hospitalier Régional, Orléans
  - Arcagy-Gineco, Paris
  - Centre Hospitalier Lyon-sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - ICO René Gauducheau, Saint-Herblain
  - Hôpital Civil, Strasbourg

REFERENCES:
- [Derived] Berton D, Floquet A, Lescaut W, Baron G, Kaminsky MC, Toussaint P, Largillier R, Savoye AM, Alexandre J, Delbaldo C, Malaurie E, Barletta H, Bosacki C, Garnier-Tixidre C, Follana P, Laharie-Mineur H, Briac Levache C, Valenza B, Dechartres A, Mollon-Grange D, Selle F. Real-World Experience of Bevacizumab as First-Line Treatment for Ovarian Cancer: The GINECO ENCOURAGE Cohort of 468 French Patients. Front Pharmacol. 2021 Sep 20;12:711813. doi: 10.3389/fphar.2021.711813. eCollection 2021. PMID 34616296